CLINICAL TRIAL: NCT04465045
Title: Unexplained Infertility Treated by Hysteroscopy-laparoscopy : Predictive Factors of Pregnancy
Brief Title: Unexplained Infertility Treated by Hysteroscopy-laparoscopy
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0084
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Unexplained Infertility
Keywords: Ovulation; semen analysis; tubal patency; pelvic ultrasound scan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — some endometrial biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Unique cohort: All women, 18 to 43 years, operated from laparoscopy-hysteroscopy for unexplained infertility in montpellier university hospital
  Interventions: Procedure: Laparoscopy-hysteroscopy

INTERVENTIONS:
Procedure: Laparoscopy-hysteroscopy — Under general anesthesia, we start by a first look in laparoscopy, to look for endometriosis mainly, tubal infertility, ovarian cysts or any abnormalities that may not have been suspected on the first exam. Then we check tubal patency after a look at the uterine cavity by hysteroscopy. Then we treat everything possible to treat to improve fertility, spontaneous or with ART.

SUMMARY:
Retrospective study, including patients from january 2013 to december 2018, who were diagnosed with unexplained infertility : spontaneously ovulating women with normal pelvic ultrasound scan, patent tubes on hysterosalpingography and normal pelvic exam or pelvic MRI normal. Semen analyses were normal according to the World Health Organization criteria. Couples were referred for diagnostic laparoscopy and hysteroscopy. They were then addressed for spontaneous fertility or ART to conceive. The investigators would like to see how many surgeries were useful to assess a diagnostic, and if operating allows a satisfying pregnancy rate. The investigators would like to assess how many diagnosis was done after surgery and how many pregnancy were obtained. The investigators search other prognostic factors than age or parity.

ELIGIBILITY:
Inclusion criteria:

* 18-43y
* unexplained infertility
* operated from laparoscopy-hysteroscopy at montpellier university hospital

Exclusion criteria:

* an IMR that diagnoses formelly an endometriosis, or endometriosic ovarian cysts
* any non respect to inclusion criterias
* non respect of our definition of unexplained infertility (such as bilateral tubal issue on hysterosalpingograms)

Ages: 18 Years to 43 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: In Montpellier University center only, France : from january 2013 to december 2018 unexplained infertile couple, trying to conceive for more than one year and operated by laparoscopy-hysteroscopy
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate | 1 day
  pregnancy with an hearbeat on a pelvic ultrasound scan

SECONDARY OUTCOMES:
Number of Participants with miscarriage | 1 day
  Number of Participants with miscarriage : positive pregnancy blood test, resulting in bleeding
live birth rate | 1 day
  live birth rate : birth of a viable foetus after 24 SA
Number of Participants with fœtal losses | 1 day
  Number of Participants with Foetal losses : loss of a non viable foetus, before 24 SA
Number of Participants with ectopic pregnancy | 1 day
  Number of Participants with ectopic pregnancy: tubal pregnancy highly suspected by blood test or seen on a pelvic ultrasound scan
Number of Participants with surgical complications | 1 day
  Number of Participants withSurgical complications : during surgery, and a few days after surgery
Number of Participants with type of surgery | 1 day
  Number of Participants with type of surgery: tubal surgeries, adhesiolysis, endometriosis surgeries, hysteroscopic gestures.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Vincens, doctor of medecine, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC